CLINICAL TRIAL: NCT01670526
Title: Rivastigmine Patch in Veterans With Cognitive Impairment Following TBI
Acronym: RIVET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-003-10S; CCTA#0001 (Other: VA)
Record Dates: First submitted 2012-08-01; First posted 2012-08-22 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Traumatic Brain Injury; Cognitive Impairment
Keywords: Traumatic Brain Injury; Cognitive Impairment; Rivastigmine; Pharmacologic Actions; TBI; Memory; Cholinesterase Inhibitors; Cognition; Head Trauma
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction; Craniocerebral Trauma | interventions — Cholinesterase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivastigmine (Experimental): Rivastigmine transdermal patch
  Interventions: Drug: Rivastigmine Transdermal Patch
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Rivastigmine Transdermal Patch

INTERVENTIONS:
Drug: Rivastigmine Transdermal Patch — Cholinesterase Inhibitor
  Other Names: Cholinesterase Inhibitor

SUMMARY:
Difficulties with intellectual functioning, particularly memory functions, are common and source of long-term disability after Traumatic Brain Injury (TBI). However, there is very little information about pharmacologic (i.e., medication) treatments targeting these deficits. There are growing data showing brain abnormalities in acetylcholine, the chemical system that manages memory, in TBI. These findings provide the rationale for the use of cholinesterase inhibitors, medications that modulate this system, in TBI patients. As the prevalence of TBI among Veterans of recent military conflicts increases, becoming a "signature injury" of the Iraq and Afghanistan conflicts, it is of utmost importance to the Veterans Health Administration to collect scientific data on the efficacy of pharmacological treatments for intellectual difficulties in TBI patients. This study will evaluate the effects of the cholinesterase inhibitor rivastigmine transdermal patch in Veterans with TBI and posttraumatic memory problems. Results will provide much needed data that will help treat Veterans with TBI.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) represents one of the most significant health risks related to military duty; rapidly becoming the "signature injury" of the Iraq and Afghanistan conflicts. TBI patients often experience multiple cognitive problems, with disturbances in memory, attention, and executive functions among the most common. Disturbances in memory as well as attention are particularly problematic, as disruption of these relatively basic cognitive functions may exacerbate or cause additional disturbances in executive function, communication and other more complex cognitive domains. These cognitive deficits, especially when memory is affected, significantly impact day-to-day functioning and are the source of lingering disability and distress to the affected individuals. However, despite advances made in TBI care, treatment of cognitive deficits in TBI lag behind, forcing clinicians to provide treatment without the guidance of evidence-based scientific data. This proposal aims to begin the process of providing clinicians with evidence-based guidelines for pharmacological management of Veterans with TBI suffering from persistent cognitive deficits following their injuries. This aim will be accomplished by conducting a clinical trial in Veterans suffering from moderate to severe posttraumatic memory impairment following TBI. Specifically, this proposal will evaluate the efficacy and safety of rivastigmine transdermal patch, an intermediate-acting cholinesterase inhibitor, in this population.

The investigators hypothesize that rivastigmine transdermal patch will be more effective than, and equally safe as, placebo in the treatment of moderate to severe posttraumatic memory impairment in Veterans with TBI when tested in a randomized, multi-site, parallel design, placebo-controlled trial, at a 12-week endpoint. The exploratory hypothesis states that compared to placebo, rivastigmine patch will be more effective and equally safe in the treatment of patients who will continue in a randomized, placebo-controlled phase for a total of 26 weeks. To test these hypotheses we will evaluate the effect and the safety of rivastigmine 9.5 mg/24 hours (10cm2) transdermal patch in 138 Veterans who meet or exceed the criteria for closed, non-penetrating, mild TBI and who present at baseline with moderate to severe memory impairment. Memory impairment will be defined as a Total Recall index (Trials 1-3) of the Hopkins Verbal Learning Test-Revised (HVLT-R) that is at least 25% lower than the intelligence-adjusted expected score, as assessed by the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Information and Vocabulary subtests. The study consists of a screening period, one-week single-blind, placebo run-in phase, and a 12-week double-blind acute treatment phase (Phase I). Subjects will be randomized 1:1 to rivastigmine transdermal patch 9.5mg/24 hours (10cm2) or matching placebo. During Phase I, there will be an initial 4-week titration period followed by an 8-week continuation phase. Following the 12-week acute treatment phase, randomized patients will continue in the double-blind phase (Phase II) for additional 14 weeks or until study treatment period ends. Recruitment stage ended 2.25.16. Efficacy will be determined by comparing the proportion of patients in each treatment group who are classified as responders at week 12. Secondary measure of functional capacity assessing the impact of memory improvement on real-world functioning, other measures of cognitive domains affected in TBI, namely attention, working and episodic memory and executive functions, as well as measures of mood and quality of life will be examined. Study findings will contribute to the body of evidence needed to establish standards of care for Veterans with posttraumatic memory impairment and other cognitive deficits.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or a female of any race
* Be outpatient Veterans residing in the community
* Be 19-65 years old at the time of inclusion
* Female patients of childbearing potential must have a negative pregnancy test at baseline and must practice an acceptable method of birth control during the trial
* Satisfy the following diagnostic criteria:

  * A history of previous head trauma(s) at least 12 months prior to study enrollment as determined by TBI diagnostic assessment
  * Closed head injury (non-penetrating) based on International Classification of Disease (ICD) 9 CM (Clinical Modification) 10 diagnosis code 854.0 as determined by TBI diagnostic assessment
  * Meet or exceed the modified American Congress of Rehabilitation Medicines (ACRM) criteria for Mild TBI as determined by TBI diagnostic assessment
* Have a deficit in the area of verbal memory
* Have subjective memory impairment that was reported to be present from the time of injury or shortly thereafter to be associated with brain injury
* Satisfy the Diagnostic and Statistical Manual (DSM, 4th edition) for cognitive disorder not otherwise specified, dementia due to TBI, or amnestic disorder due to TBI
* Demonstrate willingness to accept randomization
* Provide written informed consent to participate in the study

Exclusion Criteria:

* Have a medical condition that can interfere with the diagnostic process and the assessment of clinical and mental status, or possibly endanger their health. Such conditions include, but are not limited to endocrinological, neurological (including epilepsy), cardiovascular (including clinically significant bradyarrhythmia, resting heart rate <50 without a pacemaker or treating physician's approval), pulmonary, hematologic, hepatic, and renal conditions, and significant laboratory abnormalities as determined by Study Chair.
* Have a current diagnosis of any primary neurodegenerative disorder, including Huntington's disease, Parkinson's disease, or DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision) dementia (other than Dementia Due to Head Trauma).
* Have suicidal ideations or have been judged to be a significant suicide risk per clinical judgment and the Columbia Suicide Severity Rating Scale (C-SSRS).
* Have a history of DSM-IV-TR substance (drug and/or alcohol) dependence disorder within the last 5 years or a history of a substance abuse disorder within the past 6 months.
* Have a DSM-IV-TR lifetime and current psychotic disorder (except lifetime depression with psychotic features), bipolar disorder, or pre-TBI onset attention-deficit/hyperactivity disorder.
* Have current PTSD symptoms that can bias or interfere with cognitive and clinical assessments as determined by study site PI.
* Have demonstrated suboptimal effort on cognitive testing as defined by:

  1. Test of Memory Malingering (TOMM) raw score below 45 on either Trial 2 or the Retention Trial, or
  2. Green's Medical Symptom Validity Test (MSVT) score of 85% on any one of the Immediate Recall, Delayed Recall, or Consistency indices.
* Have demonstrated a lack of tolerability to rivastigmine treatment in the past or severe reactions to other cholinesterase inhibitors as determined by the site investigator.
* Be taking medications that significantly affect cognitive functioning in TBI population and/or may enhance the beneficial/adverse/toxic effect of rivastigmine or vice versa. These compounds include, but are not limited to, centrally-acting anticholinergic drugs (e.g., atropine), other cholinesterase inhibitors (e.g., donepezil, galantamine), and agents that augment cerebral catecholaminergic function (e.g., psychostimulants, amantadine, memantine, selegiline, levodopa, etc). Subjects receiving modafinil may be considered for inclusion if they have been on a stable dose for a minimum of 3 months, and if all inclusion criteria are met. Treatment of non-exclusionary comorbid psychiatric symptoms with compounds that include, but are not limited to, antidepressants, anxiolytics, sedative-hypnotics, anticonvulsants, and atypical antipsychotics will be permitted provided that: 1) the site investigator, based on review of medical history, records, and current medications and in consultation with the Study Chair, concludes that the agent(s) are neither cause(s) of nor significant contributor(s) to the potential subject's memory impairment; 2) the dose of the agent(s) has been stable for the 3 months preceding study participation; and 3) the dose of the agent(s) remains stable, where clinically feasible, throughout the study. For medications prescribed for non-exclusionary conditions on as needed basis, particularly when those medications include benzodiazepines, sympathomimetics, antitussive agents or potentially sedating analgesics - every use will be documented by the subject and will not be taken within 24 hours of performing study-related cognitive testing. (Appendix A: Exclusionary Medications).
* Have been exposed to other cholinesterase inhibitors in the 30 days prior to randomization.
* Have a history of penetrating brain injury, cerebrovascular disease, cerebral neoplasm, major brain surgery, or multiple sclerosis.
* Have a significant visual or auditory deficit that may interfere with ability to complete study assessments.
* Have a limited ability to speak and read English.
* Be participating in another clinical trial with active intervention.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Brawman-Mintzer, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (8):
- United States (8):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Lincoln Community-Based Outpatient Clinic, Lincoln, NE, Lincoln, Nebraska
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brody DL. Taking a Bite of the Elephant: A Well-Executed Clinical Trial Answers a Key Question About Rivastigmine Treatment for Memory Impairment after TBI. J Neurotrauma. 2021 Jul 15;38(14):1889. doi: 10.1089/neu.2021.29110.editorial. No abstract available. PMID 34213962
- [Derived] Brawman-Mintzer O, Tang XC, Bizien M, Harvey PD, Horner MD, Arciniegas DB, Raskind M, Johnson-Greene L, Martineau RJ, Hamner M, Rodriguez-Suarez M, Jorge RE, McGarity S, Wortzel HS, Wei Y, Sindowski T, Mintzer J, Kindy AZ, Donovan K, Reda D. Rivastigmine Transdermal Patch Treatment for Moderate to Severe Cognitive Impairment in Veterans with Traumatic Brain Injury (RiVET Study): A Randomized Clinical Trial. J Neurotrauma. 2021 Jul 15;38(14):1943-1952. doi: 10.1089/neu.2020.7146. Epub 2021 Mar 8. PMID 33514274
- See also: The War Related Illness and Injury Study Center offers services for combat veterans — http://www.warrelatedillness.va.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rivastigmine | Placebo
Started | 49 | 45
Completed | 37 | 39
Not Completed | 12 | 6
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivastigmine | Placebo | Total
Number analyzed (Participants) | 49 | 45 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 45 | 94
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 47 | 43 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 30 | 34 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 49 | 45 | 94

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Demonstrated Improvement From Baseline on the Hopkins Verbal Learning Test-Revised (HVLT-R) Total Recall
Description: The primary efficacy measure was the Hopkins Verbal Learning Test - Revised (HVLT-R) Total Recall Index. HVLT-R was administered at screen, baseline, weeks 4, and 12. The HVLT is a measure that assesses verbal learning and memory. Alternate versions of the HVLT-R were administered at each of the different time points. The test consists of 12 words which are read to participants for three consecutive trials, each trial followed by free recall. The Total Recall score is the total number of words recalled over the three trials. The primary endpoint evaluation was to compare the proportion of patients who demonstrated improvement from baseline on the HVLT-R Total Recall of at least 5-word and at week 12 between the treatment and placebo group.
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Rivastigmine | Placebo
Number analyzed (Participants) | 49 | 45
Participants | 20 | 23

2. Secondary Outcome: Twelve-week Change in University of California San Diego Performance-based Skills Assessment - Brief (UPSA-B)
Description: UPSA-B is a validated performance-based measure to evaluate the impact of rivastigmine-mediated memory improvements on the ability to perform tasks required for day-to-day functioning in two subdomains of financial management and communication. The scale goes from (0-100) and high score indicates better functions. Comparison of difference in mean changes of UPSA-B from baseline to 12-week follow-up between two groups.
Time Frame: 12 weeks
Population: Participants complete 12 weeks follow up included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine | Placebo
Number analyzed (Participants) | 49 | 45
units on a scale | -0.9 (6.4) | 3.3 (8.5)

3. Secondary Outcome: Twelve-week Change in The PTSD Symptom Checklist-Military Version (PCL-M)
Description: PCL-M is a validated 17-item self-report measure of DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision) symptoms of PTSD.The PCL-M asks about problems in response to "stressful military experiences." Items are rated on a 5-point scale ranging from 1 ("not at all") to 5 ("extremely"). Higher score indicates more stressful.
  Comparison of difference in mean changes of PCL-M from baseline to 12-week follow-up between two groups.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine | Placebo
Number analyzed (Participants) | 49 | 45
units on a scale | -1.4 (8.9) | -4.4 (9.8)

4. Secondary Outcome: Twelve-week Change in Beck Depression Inventory-II (BDI-II)
Description: Beck Depression Inventory-II (BDI-II) is a validated 21-question multiple-choice self-report inventory, one of the most widely used instruments for measuring the severity of depressive symptoms. Each answer is scored on a scale value of 0 to 3. Higher score indicates more severe depression.
  To compare the differences in mean changes of BDI-II between two groups using two groups from baseline to week 12.
Time Frame: 12 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine | Placebo
Number analyzed (Participants) | 49 | 45
units on a scale | -1.4 (8.8) | -0.7 (9.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected on study participants starting from when the first participant was enrolled, December 29, 2012 through June 16, 2016 (3 1/2 years).
Description: Adverse event (AE) and serious adverse event (SAE) data based on system organ classes and preferred terms which are derived from MedDRA (Medical Dictionary for Regulatory Activities) coding. MedDRA terminology is the international medical terminology developed under the auspices of the International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH).
Arm/Group | Rivastigmine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/45
Serious Adverse Events (participants affected / at risk) | 4/49 | 4/45
Other Adverse Events (participants affected / at risk) | 10/49 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivastigmine (N=49) | Placebo (N=45)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
post traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
self serious ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Somnolence (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivastigmine (N=49) | Placebo (N=45)
accident at work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — work injury, non study related
Application site erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
application site irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Application site pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Carpel tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Knee operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nauseau (Gastrointestinal disorders) | 1 (1) | 0 (0)
Product adhesion issue (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No